CLINICAL TRIAL: NCT03788694
Title: Pilot Study of Open Label, Intranasal Ketamine for Suicidal Ideation in Veterans
Brief Title: Intranasal Ketamine for Suicidal Ideation in Veterans
Status: Withdrawn | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Study was never funded nor started, no participants were enrolled
Sponsor: Bronx Veterans Medical Research Foundation, Inc (Other)
Collaborators: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Principal Investigator, Marianne Goodman, Associate Director, VISN 2 Mental Illness, Reseach, Education, Clinical Center (MIRECC) Director, Suicide Prevention and Treatment Research Program, James J. Peters Veterans Affairs Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GOO-17-048
Record Dates: First submitted 2018-12-26; First posted 2018-12-27 (Actual); Last update posted 2023-08-07 (Actual); Status verified 2023-08

CONDITIONS: Suicidal Ideation
Keywords: Ketamine; Veteran; Suicide; Suicidal Ideation
MeSH Terms: conditions — Suicidal Ideation; Suicide | interventions — Ketamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Intranasal Ketamine (Experimental): Subjects will receive study medication, intranasal ketamine.
  Interventions: Drug: Ketamine

INTERVENTIONS:
Drug: Ketamine — 8 doses of intranasal ketamine; 40 mg per dose.

SUMMARY:
The objective of the current study is to investigate the safety, efficacy, and feasibility of multiple doses of intranasal (IN) ketamine for suicidal ideation Veterans.

DETAILED DESCRIPTION:
To address the significant need for effective treatment of suicidal ideation in Veterans, this trial is designed as an open label pilot study of intranasal ketamine in 15 people.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients, 21-70 years of age
2. Female individuals who are not of childbearing potential (i.e., surgically sterile, postmenopausal for at least one year) or using a medically accepted reliable means of contraception. Women using oral contraceptive medication for birth control must also be using a barrier contraceptive. Women of childbearing potential must also have a negative pregnancy test at screening and at pre-administration
3. Any non-psychotic disorder diagnosis
4. Score >4 on the suicide item of the Montgomery-Asberg Depression Rating Scale (MADRS-SI; range 0-6)for clinically significant suicidal ideation or past suicide attempts
5. Each participant must have a level of understanding sufficient to agree to all tests and examinations required by the protocol and must sign an informed consent document
6. Each participant must agree to avoid future enrollment in ketamine trials.

Exclusion Criteria:

1. current psychotic symptoms or lifetime history of primary psychotic disorder
2. active substance use in the preceding two weeks or needing medical attention for withdrawal
3. neurodevelopmental disorder (e.g., ASD)
4. major neurocognitive disorder (e.g., Alzheimer's type dementia)
5. serious cardiac disease
6. suicide attempt precipitating current admission requiring medical stabilization
7. Lifetime histories of autism, mental retardation, pervasive developmental disorders, or Tourette's syndrome
8. Women who are either pregnant or nursing
9. Hypertension (systolic BP >160 mm Hg or diastolic BP >90 mm Hg) at screening or immediately prior to treatment with study drug
10. Previously received ketamine for refractory depression.

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2020-01-31 (Actual); Study Completion 2020-04-30 (Actual)

PRIMARY OUTCOMES:
Change in Beck Scale for Suicidal Ideation (BSSI) | Baseline Visit to End of Treatment Visit- approximately 3-4.5 weeks
  Beck Scale is a 21-item self or clinician administered instrumentation used to measure the current intensity of patients' specific attitudes, behaviors and plans to commit suicide. Score range 0-42, with higher score indicating higher intensity.

SECONDARY OUTCOMES:
Montgomery-Asberg Depression Rating Scale (MADRS) | Baseline Visit to End of Treatment Visit- approximately 3-4.5 weeks
  The MADRS is a 10-item instrument used for the evaluation of depressive symptoms in adults and for the assessment of any changes to those symptoms. Higher MADRS score indicates more severe depression, and each item yields a score of 0 to 6. The overall score ranges from 0 to 60.
The Quick Inventory of Depressive Symptomatology, Self-Report (QIDS-SR) | Baseline Visit to End of Treatment Visit- approximately 3-4.5 weeks
  QIDS-SR is a 16-item self-rated instrument designed to assess the severity of depressive symptoms present in the past seven days (Rush et al. 2003). The 16 items cover the nine symptom domains of major depression, and are rated on a scale of 0-3.

CONTACTS AND LOCATIONS:
Locations (1):
- James J. Peters VA Medical Center, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in publications as well as study protocol, statistical analysis plan, informed consent form.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: 6 months after publication and will remain available for 5 years.